CLINICAL TRIAL: NCT00985439
Title: A Phase 2, Randomized, Double-Blind, Single-Dose, Parallel-Group, Active- and Placebo-Controlled Study of Diclofenac [Test] Capsules for the Treatment of Pain After Surgical Removal of Impacted Third Molars
Brief Title: Study of Diclofenac Capsules to Treat Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIC2-08-03
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-03

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diclofenac Test (lower dose) (Experimental): One 18-mg Diclofenac Test Capsule and 1 placebo capsule
  Interventions: Drug: Diclofenac Test (lower dose)
- Diclofenac Test (upper dose) (Experimental): One 35-mg Diclofenac Test Capsule and 1 placebo capsule
  Interventions: Drug: Diclofenac Test (upper dose)
- Celecoxib 400 mg (Active Comparator)
  Interventions: Drug: Celecoxib 400 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Test (lower dose) — 18-mg Single dose
  Arms: Diclofenac Test (lower dose)
Drug: Diclofenac Test (upper dose) — 35-mg Single dose
  Arms: Diclofenac Test (upper dose)
Drug: Celecoxib 400 mg — Capsules 2 x 200 mg Single-dose
  Arms: Celecoxib 400 mg
Drug: Placebo — Capsules 2 Single-dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Diclofenac Test Formulation Capsules are safe and effective for the treatment of dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 50 years of age
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Patient requires extraction of 2 or more third molars
* Patient must be willing to stay at the study site overnight

Exclusion Criteria:

* Patient has hypersensitivity, allergy, or clinically significant intolerance to any medications to be used in the study, or related drugs
* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen or alcohol breathalyzer test
* Patient has taken another investigational drug within 30 days prior to Screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Premier Research Group Limited, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Celecoxib 400 mg | Placebo
Started | 49 | 51 | 51 | 51
Completed | 49 | 51 | 50 | 51
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Celecoxib 400 mg | Placebo | Total
Number analyzed (Participants) | 49 | 51 | 51 | 51 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 51 | 51 | 51 | 202
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.1 (5.10) | 22.3 (4.58) | 22.7 (3.30) | 22.6 (4.22) | 22.4 (4.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 34 | 25 | 116
  Male | 22 | 21 | 17 | 26 | 86
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 51 | 51 | 202

OUTCOME MEASURES:

1. Primary Outcome: Total Patient Pain Relief Over 0 to 12 Hours.
Description: Total patient pain relief was assessed as a time-weighted sum of the patient pain assessments at each individual time point from 0-12 hours.
  Values for TOTPAR are measured from 0 to 4 on the Pain Relief Scale 0 None Min; 1 A little; 2 Some; 3 A lot; 4 Complete Max
  The TOTPAR is a weighted measure of the observations; the minimum possible value is 0 and the maximum possible value is 60.
Time Frame: 12 hours.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Diclofenac Test (Lower Dose): 18-mg
- Diclofenac Test (Upper Dose): 35-mg
Arm/Group | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Celecoxib 400 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 51 | 51
units on a scale | 17.770 (13.7607) [14.020 to 21.520] | 16.893 (12.7634) [13.215 to 20.571] | 14.685 (15.0524) [11.008 to 18.363] | 5.486 (11.5272) [1.802 to 9.170]
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 11.407, 95% CI 2-sided [6.195 to 16.619], Standard Error of Mean 2.6430

ADVERSE EVENTS:
Arm/Group | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Celecoxib 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 27/49 | 31/51 | 32/51 | 27/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Test (Lower Dose) (N=49) | Diclofenac Test (Upper Dose) (N=51) | Celecoxib 400 mg (N=51) | Placebo (N=51)
Alveolar Osteitis (Gastrointestinal disorders) | 0 | 0 | 3 | 4
Dizziness (Nervous system disorders) | 3 | 4 | 3 | 6
Ear Pain (Ear and labyrinth disorders) | 3 | 1 | 2 | 1
Headache (Nervous system disorders) | 7 | 14 | 9 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 6 | 9 | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 12 | 11 | 10 | 9
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No